CLINICAL TRIAL: NCT04158102
Title: A Phase 1, Open Label Study to Evaluate the Pharmacokinetics and Safety of EXPAREL® Following Subcutaneous Administration in Healthy Chinese Subjects
Brief Title: Evaluate the Pharmacokinetics and Safety of EXPAREL® Following Subcutaneous Administration in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nuance Pharma (shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NB-EXP-1001
Record Dates: First submitted 2019-11-05; First posted 2019-11-08 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-11

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 20 mg single dose cohort (Experimental): Subjects would receive a 20 mg single dose of EXPAREL®
  Interventions: Drug: Bupivacaine liposome injectable suspension

INTERVENTIONS:
Drug: Bupivacaine liposome injectable suspension — Single dose of Bupivacaine liposome injectable suspension 266 mg in 20 mL
  Other Names: EXPAREL®

SUMMARY:
This is a single-center, open-label, single-dose study to evaluate the safety, pharmacokinetics in healthy subjects

DETAILED DESCRIPTION:
This is a phase I, open-label, single-dose in healthy subjects conducted at single center.The objectives are to evaluate the metabolic and safety profile of EXPAREL®. Each volunteer will receive one dose of the investigational drug via subcutaneous injection at multiple points during the study period. Study duration is around 54 days, including screening, confinement, ambulatory visit and a phone follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese male or female subjects, and his/her biological parents and grandparents are of Chinese ethnicity.
2. Aged ≥18 and ≤55 years of age at screening, inclusive.
3. Willing and able to give written informed consent and comply with the study visit schedule, study procedures and restrictions.
4. Generally, in good health with no clinically significant abnormalities as determined by medical history, physical examination, 12-lead ECG and clinical laboratory tests.
5. Have a body mass index (BMI) between 19.0 and 24.0 kg/m2, inclusive, and a body weight ≥50 kg at screening visit and baseline visit (Day -1).

Exclusion Criteria:

1. Female subjects who are pregnant (positive pregnancy result at screening and on Day -1), or lactating.
2. Female subjects of child bearing potential and sexually active don't agree to use medically acceptable contraceptive (e.g. insertable, injectable, transdermal, hormonal contraceptive) from the date of consent given until 30 days after administration of study drug. Menopausal woman don't have her menopausal status confirmed by follicle-stimulating hormone test at screening.
3. Male subjects who are sexually active don't agree to use condom plus spermicide since the dosing day till 90 days after administration of study drug.
4. Male subjects don't agree not to donate sperm since the dosing day till 90 days after administration of study drug.
5. Presence of any concomitant clinically significant diseases, that would interfere with the study based on the investigator's discretion.
6. History of hypersensitivity or idiopathic reaction to amide-type local anesthetics.
7. Has a positive urine drug screen result for drugs of abuse or a positive blood alcohol test at the Screening Visit or baseline visit (Day-1).
8. Has an abnormal (clinically significant) ECG at the screening visit. Entry of any subject with an abnormal (but not clinically significant) ECG must be approved and documented by signature of the Investigator or medically qualified subinvestigator.
9. Has a supine BP outside the ranges of 90 to 140 mmHg for systolic BP and 50 to 90 mmHg, inclusive, for diastolic BP, or resting pulse rate outside the range of 40 to 100 beats per minute. If any of the values are out of range, the assessment may be repeated twice for eligibility determination at the screening visit or baseline visit (Day-1).
10. Positive HIV test result at screening.
11. Positive testing for HBs Antigen and/or a positive Hepatitis C antibody test result at screening.
12. Has an abnormal laboratory values outside the reference range that are of clinical significance which may suggest of an underlying disease such as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values, greater than 1.5 times the upper limit of normal.
13. Intake prescription or over the counter products (vitamins, dietary supplements, herbal preparations, etc.) within 14 days or less than 5 half-lives (whichever is longer) prior to screening visit.
14. Blood loss or donation more than 450ml within 3 months prior to dosing.
15. Previous participation in an EXPAREL® study.
16. Administration of an investigational drug within 30 days or 5 elimination half-lives of the investigational drug, whichever is longer, prior to study drug administration, or planned administration of another investigational product or procedure during the subject's participation in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
plasma concentration | up to 14 days
  Maximum observed plasma concentration (Cmax)
Area under the plasma concentration-versus-time curve | up to 14 days
  Area under the plasma concentration-versus-time curve from time 0 extrapolated to infinity after drug administration (AUC0-∞)

SECONDARY OUTCOMES:
Incidence of adverse events（AEs）which are related to exparel injection | up to 21 days
  Adverse events refer to any treatment related abnormality with clinical significance identified by means of vital signs examination, physical check-up, twelve leads electrocardiogram inspection and laboratory tests throughout the study. Adverse events reported by subjects would also be recorded in the entire trial. All these abnormal cases described above would be reported as incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Cheung, Doctor, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- HUK Phase 1 clinical trials center, Hong Kong, Hongkong, China

REFERENCES:
- [Derived] Cheung BM, Ng PY, Liu Y, Zhou M, Yu V, Yang J, Wang NQ. Pharmacokinetics and safety of liposomal bupivacaine after local infiltration in healthy Chinese adults: a phase 1 study. BMC Anesthesiol. 2021 Jul 27;21(1):197. doi: 10.1186/s12871-021-01407-5. PMID 34315419